CLINICAL TRIAL: NCT01248039
Title: The Influence of Preoperative Pain, Function, and Activity on Time to Fulfill Discharge Criteria for Total Hip and Knee Arthroplasty Patients
Brief Title: Preoperative Pain, Function, and Activity for Total Hip and Knee Arthroplasty Patients
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Bente Holm, Physiotherapist for development and research, Hvidovre University Hospital
Other Study IDs: H-4-2010-FSP2; PRE-THA-TKA (Registry Identifier: H-4-2010-FSP2)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Arthroplasty
Keywords: Muscle strength, functional performance, joint replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total arthroplasty: Patients with osteoarthrosis going for hip or knee arthroplasty

SUMMARY:
This study wish to show if the preoperative level of pain, function or activity for hip and knee arthroplasty patients has any predictive value of the time it takes to fulfill the well-defined discharge criteria.

DETAILED DESCRIPTION:
The investigators would like to be able to identify those patients, for whom it will take longest time to fulfill the discharge criteria. With this knowledge the investigators will be able to initiate sufficient treatment already before operation.

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty patients
* Total knee arthroplasty patients

Exclusion Criteria:

* Inability to speak and understand Danish
* Inability to perform the functional measurements due to other conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Concesutive hip and knee arthroplasty patients from a department of orthopaedic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Leg muscles strength | 7 months
  Maximal muscle force tested for one leg at a time in a Power Rig Mashine

SECONDARY OUTCOMES:
Functional performance | 7 months
  Tested by: Timed Up & Go test, 10 meter fast speed walking test

CONTACTS AND LOCATIONS:
Overall Officials: Bente Holm, MSc, Principal Investigator — The Lundbeckcenter for hip and knee surgery, University Hospital at Hvidovre, Kettegaard Allé 30, DK-2650 hvidovre, Denmark
Locations (1):
- Department of Surgery, Univerity Hospital at Hvidovre, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Holm B, Bandholm T, Lunn TH, Husted H, Aalund PK, Hansen TB, Kehlet H. Role of preoperative pain, muscle function, and activity level in discharge readiness after fast-track hip and knee arthroplasty. Acta Orthop. 2014 Sep;85(5):488-92. doi: 10.3109/17453674.2014.934186. Epub 2014 Jun 23. PMID 24954491